CLINICAL TRIAL: NCT00921141
Title: Assessment of Complications, Quality of Life and Easiness of Use of Implantable Central Venous Access Ports : Cohort and Prospective Study
Brief Title: Assessment of Complications, Quality of Life and Easiness of Use of Implantable Central Venous Access Ports
Acronym: CCI
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: CCI; CCI
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: Implantable central venous access ports, cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study population: Patient with cancer requiring a long-term central venous catheter

SUMMARY:
This is a prospective, descriptive and observational study of the anticancer center practice

ELIGIBILITY:
Inclusion Criteria:

* Patient with any cancer, requiring a central venous catheter
* No contraindication for any surgery with local or complete anaesthesia

Exclusion Criteria:

* Previous Xylocaine or Lidocaine allergy
* Clinic superior vena cava syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients requiring the implementation of a catheter in an anticancerous center
Sampling Method: Non-Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Incidence and collection of complications for the patients requiring an implantable central venous access ports substitution/change | Until the implantable central venous access ports removal

SECONDARY OUTCOMES:
Brief description of the different risk factor for morbidity | Until the implantable central venous access ports removal
Assessment of the implantable central venous access ports ease-of-use for nurses according to the modalities of implementation and patient features | Until the implantable central venous access ports removal
Assessment of the patient quality of life | Before central venous access ports implementation, at the first day of chemotherapy, and during the cycle 4 of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice NARDUCCI, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France